CLINICAL TRIAL: NCT06971666
Title: Relationship Between Dietary Inflammatory Potential, Markers of Inflammation, Microbiota and Risk of Anxiety and Depression in Young People With Obesity
Brief Title: Dietary Inflammatory Potential in Young Pleople With Obesity
Acronym: DIP
Status: Not yet recruiting | Type: Observational
Sponsor: Instituto Tecnológico y de Estudios Superiores de Occidente (Other)
Responsible Party: Sponsor
Other Study IDs: ITESO-DIP-2025
Record Dates: First submitted 2025-01-20; First posted 2025-05-14 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Obesity; Dietary Inflammatory Index (DII)
Keywords: obesity; dietary inflammatory potential; dietary inflammatory index; inflammatory markers; gut microbiota; anxiety; depression
MeSH Terms: conditions — Obesity; Anxiety Disorders; Depression

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Observational, cross-sectional, analytical, and correlational: An observational, cross-sectional, analytical, and correlational study will be conducted on young individuals with obesity, diagnosed with Body Mass Index (BMI). The study aims to analyze the correlation between Dietary inflammatory potential (DIP), inflammatory markers, intestinal dysbiosis, exercise patterns, and the risk of anxiety and depression

SUMMARY:
The increase in adipose tissue in the young population is one of the most important and worrying public health problems because it persists in adulthood, constituting a risk factor for chronic degenerative diseases with social, economic, and environmental effects. The etiology of obesity is multifactorial and is associated with a low-intensity chronic inflammation process. Therefore, side effects of the digestive, nervous, endocrine, and immunological levels are closely related. Thus, understanding the impact of dietary components on the immune response and the pathophysiological complications of obesity will strengthen information on nutritional patterns with lower inflammatory implications.

DETAILED DESCRIPTION:
1. Background

   Obesity has become one of the most critical challenges in public health. It has become a global epidemic due to the exponential growth of obesity over the last 30 years, affecting developed and developing countries with a notable impact on the latter. In Mexico, the combined prevalence of overweight and obesity in adults is 75.2%, of which 36.9% correspond precisely to the prevalence of obesity.

   This pathology has a multifactorial etiology, links lifestyle, environment, and genetics, and is modulated by multiple interactions between psychological, cultural, and physiological factors. The World Health Organization defines obesity as the abnormal or excessive accumulation of adipose tissue, which can harm health. This accumulation of triglycerides in the adipocyte alters the secretion of specific molecules of the immune system, which causes a cascade of inflammation mediated by the secretion of inflammatory molecules.

   Likewise, it is observed that obese subjects present intestinal dysbiosis that leads to intestinal permeability that allows the passage of lipopolysaccharides from Gram-negative bacteria into the bloodstream. There, they are recognized as toxic agents by the immune system, and the secretion of inflammatory cytokines occurs. The immune response derived from increased adipose tissue and intestinal dysbiosis compromises different brain regions involved in regulating behavior, eating patterns, perception of satiety, and being involved in cognition and mood related to physical inactivity and more significant weight gain. The continuous circulation of inflammatory cytokines and their accumulation in organs, including the central nervous system, is a risk factor for altering neurotransmitters and signal transduction that could result in depression.

   In addition to the above, a close relationship has been reported between diet and the regulation of the inflammatory response, so changes in the dietary patterns of the Mexican population could be directly related not only to the excessive accumulation of adipose tissue but also to the persistent inflammatory response in this pathology. The Dietary Inflammatory Potential (DIP) tool has been used to evaluate the inflammation caused by an individual's diet based on their dietary inflammatory index (DII). The DII allows us to associate foods and their nutrients with markers that show pro-inflammatory or anti-inflammatory processes.

   Studies have analyzed the association of DIP with different diseases, such as vascular diseases, cancer, metabolic syndrome, and dysbiosis in patients with constipation. However, in the literature, three publications are identified that analyze DIP in people with obesity, where they consider that subjects with this disease already start from an inflammatory process. These studies evaluate this relationship between 20 and 60 years, which represents an extensive range of the population and implies a series of possible analysis biases inherent to the different age groups included in the sample and their metabolic and immunological particularities. It also stands out that none of these studies have been carried out in Mexico.
2. General objective

   To evaluate the relationship between Dietary Inflammatory Potential, markers of inflammation, microbiota, and risk of anxiety and depression in young people with obesity.
3. Hypothesis

   There is a relationship between Dietary Inflammatory Potential, inflammation markers, microbiota, risk of anxiety, and depression in young people with obesity.
4. Methodology

An original observational, cross-sectional, analytical, and correlational study in young people with obesity diagnosed with Body Mass Index. As part of the techniques and procedures, height and weight will be measured using the ISAK methodology to obtain the body mass index (BMI) and body mass with Dual X-ray Densitometry. Meanwhile, changes in intestinal microbiota and immunological parameters will be determined using the sequencing technique and ProQuantum High-Sensitivity Immunoassays, respectively. Questionnaires for evaluation of alimentary frequency, diet diversity, physical activity, and symptoms of anxiety and depression will be done.

ELIGIBILITY:
Inclusion Criteria:

* Both sexes with no gender exclusion
* Age between 18 and 24 years
* Body Mass Index (BMI) ≥ 30 kg/m²
* Signed informed consent

Exclusion Criteria:

* Pregnancy or expected pregnancy within the next month
* Women who are breastfeeding
* Diagnosed conditions such as: diabetes mellitus, hypertension, renal or hepatic insufficiency, infectious diseases, inflammatory diseases, or any neoplastic disease
* Conditions with dietary restrictions, such as celiac disease or history of gastric bypass surgery
* Active alcoholism with a daily intake exceeding 50 g/day
* Significant anticipated changes in diet or exercise within 15 days prior to the study's start
* History of drug or medication abuse
* Eating disorders
* Participation in any study involving investigational products within the 3 months prior to the start of the study
* Treatment with anti-inflammatory drugs, antibiotics, and/or antidepressants in the month prior to the study's start
* Consumption of nutraceuticals containing prebiotics, probiotics, or immunomodulators within 15 days prior to the study's start
* Individuals who choose to discontinue participation after the data collection process has started.
* Individuals who do not consent to the collection of any of the required samples (blood, diet, or stool) during the data collection phase.

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Individuals aged 18 to 24 years, diagnosed with obesity based on Body Mass Index (BMI), recruited from the Centro Universitario de Tonalá at the University of Guadalajara and ITESO between August 2024 and June 2025, residing in the Guadalajara Metropolitan Area.
Sampling Method: Non-Probability Sample
Enrollment: 170 (Estimated)
Dates: Start 2025-06-20 (Estimated); Primary Completion 2026-11-22 (Estimated); Study Completion 2027-01-07 (Estimated)

PRIMARY OUTCOMES:
Dietary Assessment | 1.5 years
  Dietary intake will be estimated from a validated semiquantitative food frequency questionnaire (FFQ) that represents food consumption for the last 12 months. For each item, regular portion size will be established, and then frequencies of consumption will be available, ranging from "never" to "6 or more times/day". Energy and nutrient intakes will be obtained by multiplying the frequency by the serving size from Mexican food composition.
Dietary Inflammatory Index, DII | 1.5 years
  For the Dietary Inflammatory index, 45 food parameters related (positively or negatively) to inflammatory markers such as IL beta, IL4, IL6, IL10, TNF alpha, and CRP will be used. The score for each dietary parameter will be multiplied by each participant's intake, resulting in a numerical score ranging from -8 to +8.
Dietary Inflammatory Potential, DIP | 1.5 years
  The DIP will be obtained by analyzing the Dietary assessment and the Dietary Inflammatory Index intake, which will then be converted to a percentile score of 2 and subtracted by 1. The percentile score will be multiplied by the inflammatory effect score. All food parameters sill be summed to create the score. The score will be in quartiles: Q1, highly anti-inflammatory, Q2, anti-inflammatory, Q3, inflammatory; and Q4, highly inflammatory

SECONDARY OUTCOMES:
Inflammatory markers | 1.5 years
  For the determination of IL6, IL1 beta, IL10, and MCP-1 markers, a blood sample will be collected and then analyzed using the high-sensitivity ProQuantum™ technique. The assay workflow with one antibody incubation step prior to placing the plate in qPCR to determine levels of protein in picogram per milliliter, pg/mL.
C-reactive protein (CRP) | 1.5 years
  Determination of C-reactive protein levels will be determined by measuring the protein in a blood sample by visual agglutination. The results will be reported as positive or negative.
Intestinal microbiota | 1.5 years
  Analyses of intestinal microbiota will be performed by Rasmus sequencing on Illumina's MiSeq equipment. High-quality sequences will be classified into operational taxonomic units (OTUs) using the RDP database platform (Ribosomal Database Project) for the 16S rDNA gene with a bootstrap cutoff of 80%. Only OTUs representing more than 0.1% of the total sequences in each sample will be considered in subsequent statistical analyses.
Height | 1.5 years
  Height (mt) will be recorded. The technique extension requires the subject to stand with the feet apart at a 45° angle and the heels together, the posterior aspect of the buttocks, and the upper back resting on the stadiometer. The head should be in the Frankfort plane. The subject is asked to take a deep breath and hold it; the scorer places the square, triangular piece firmly over the vertex, squeezing the hair as tightly as possible. The measurement will be taken at the end of a deep breath.
Body weight | 1.5 years
  Body weight (kg) will be checked when the scale is in the zero register. Then, the subject will stand in the center of the scale without support, with the weight distributed evenly between both feet. The head should be elevated, and the eyes should look directly forward.
Body Mass Index (BMI) | 1.5 years
  The body mass index (BMI) will be calculated by dividing the weight, previously obtained from the person evaluated, by the squared height (mt). BMI will be reported in categories: <18.5, 18.5 - 24.9, 25-29.9 and >30
Dual-Energy X-Ray Absorptiometry (DXA) | 1.5 years
  For DXA, the patient will be instructed to wear non-metallic clothing and remove any metallic objects that might interfere with the procedure. Subsequently, the patient will lie on the densitometer bed. The scanner will emit a low dose of radiation (less than 0.01 mSv) to measure the density of body tissues, from which the mass (in kilograms) of various structural body tissues will be estimated.
Bioelectrical Impedance Analysis (BIA) | 1.5 years
  The patient will be instructed to wear non-metallic clothing and remove any metallic objects that might interfere with the procedure. The patient will then lie on an examination table, and electrodes from the impedance analyzer (SECA mBCA 525) will be placed on the body. The device will emit an electrical current at different frequencies to measure the subject's body reactance, resistance, and impedance. Based on these measurements, we will obtain the mass (in kilograms)
Anxiety | 1.5 years
  To assess anxiety, the Generalized Anxiety Disorder Scale (GAD-7) will be applied. The GAD-7 consists of seven items designed to evaluate generalized anxiety disorder (GAD). Responses will be classified using a 4-point Likert scale and categorized based on their occurrence over the past two weeks as follows:
  Minimal GAD (score ≤ 4) Mild GAD (score of 5-9) Moderate GAD (score of 10-14) Severe GAD (score ≥ 15). Any score ≥ 5 will be categorized as "more than minimal" generalized anxiety disorder. Additionally, any score ≥ 10 will be classified as "clinically relevant" generalized anxiety disorder symptomatically.
Depression | 1.5 years
  To evaluate depressive symptoms, the Patient Health Questionnaire (PHQ-9) will be used. The PHQ-9 is designed to detect self-reported symptoms of major depressive disorder (MDD). The questionnaire consists of nine items describing common depressive conditions, rated on a 4-point Likert scale based on their occurrence in the past two weeks
Movement behavior | 1.5 years
  To estimate levels of physical activity and sedentary behavior, the short version of the International Physical Activity Questionnaire (IPAQ) will be used. This questionnaire has been validated and previously applied to the Mexican population. The short version assesses hours and minutes of moderate and vigorous physical activity, as well as walking, performed in the last seven days for at least 10 continuous minutes.
Food security | 1.5 years
  The level of food security will be assessed at an individual level using the first eight questions of the Latin American and Caribbean Food Security Scale (ELCSA), which has been validated and specifically developed for the context of Latin America and the Caribbean. This scale refers to experiences of food insecurity related to poverty during the three months preceding the survey. To classify the level of food security, a categorization algorithm will be applied based on the number of affirmative responses, as follows:
  Food security (score = 0) Mild/low food insecurity (score of 1 to 3) Moderate food insecurity (score of 4 to 6) Severe food insecurity (score of 7 to 8)

IPD SHARING:
Plan to Share IPD: No
This is a project that involves data about patent

REFERENCES:
- [Background] Baltazar-Diaz TA, Gonzalez-Hernandez LA, Aldana-Ledesma JM, Pena-Rodriguez M, Vega-Magana AN, Zepeda-Morales ASM, Lopez-Roa RI, Del Toro-Arreola S, Martinez-Lopez E, Salazar-Montes AM, Bueno-Topete MR. Escherichia/Shigella, SCFAs, and Metabolic Pathways-The Triad That Orchestrates Intestinal Dysbiosis in Patients with Decompensated Alcoholic Cirrhosis from Western Mexico. Microorganisms. 2022 Jun 16;10(6):1231. doi: 10.3390/microorganisms10061231. PMID 35744749
- [Background] Hadi S, Momenan M, Cheraghpour K, Hafizi N, Pourjavidi N, Malekahmadi M, Foroughi M, Alipour M. Abdominal volume index: a predictive measure in relationship between depression/anxiety and obesity. Afr Health Sci. 2020 Mar;20(1):257-265. doi: 10.4314/ahs.v20i1.31. PMID 33402914
- [Background] Craig CL, Marshall AL, Sjostrom M, Bauman AE, Booth ML, Ainsworth BE, Pratt M, Ekelund U, Yngve A, Sallis JF, Oja P. International physical activity questionnaire: 12-country reliability and validity. Med Sci Sports Exerc. 2003 Aug;35(8):1381-95. doi: 10.1249/01.MSS.0000078924.61453.FB. PMID 12900694
- [Background] Corley J, Shivappa N, Hebert JR, Starr JM, Deary IJ. Associations between Dietary Inflammatory Index Scores and Inflammatory Biomarkers among Older Adults in the Lothian Birth Cohort 1936 Study. J Nutr Health Aging. 2019;23(7):628-636. doi: 10.1007/s12603-019-1221-y. PMID 31367727
- [Background] Cavicchia PP, Steck SE, Hurley TG, Hussey JR, Ma Y, Ockene IS, Hebert JR. A new dietary inflammatory index predicts interval changes in serum high-sensitivity C-reactive protein. J Nutr. 2009 Dec;139(12):2365-72. doi: 10.3945/jn.109.114025. Epub 2009 Oct 28. PMID 19864399
- [Background] Boutens L, Hooiveld GJ, Dhingra S, Cramer RA, Netea MG, Stienstra R. Unique metabolic activation of adipose tissue macrophages in obesity promotes inflammatory responses. Diabetologia. 2018 Apr;61(4):942-953. doi: 10.1007/s00125-017-4526-6. Epub 2018 Jan 14. PMID 29333574
- [Background] Amiri S, Behnezhad S. Obesity and anxiety symptoms: a systematic review and meta-analysis. Neuropsychiatr. 2019 Jun;33(2):72-89. doi: 10.1007/s40211-019-0302-9. Epub 2019 Feb 18. PMID 30778841
- [Background] Almeida-de-Souza J, Santos R, Barros R, Abreu S, Moreira C, Lopes L, Mota J, Moreira P. Dietary inflammatory index and inflammatory biomarkers in adolescents from LabMed physical activity study. Eur J Clin Nutr. 2018 May;72(5):710-719. doi: 10.1038/s41430-017-0013-x. Epub 2017 Dec 26. PMID 29277838